CLINICAL TRIAL: NCT06633562
Title: A Phase 1a Randomized, Double-blind, Placebo-controlled, Single Site, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of Nezavist in Healthy Adults
Brief Title: A Study to Test the Effects of Nezavist at Different Doses in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lohocla Research Corporation (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEZ-2021-01; 2R44AA024905-06 (NIH); 4R44AA024905-07 (NIH)
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Healthy; Safety Evaluation of Escalating Doses; Tolerability
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled, Single Site, Single Ascending Dose Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All research staff will be blinded to treatment given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Nezavist Cohort 1 (Active Comparator): Nezavist 500 mg in a volume of 60 mL NPO 8 hrs AM bib.
  Interventions: Drug: Nezavist SDD
- Nezavist Cohort 2 (Active Comparator): Nezavist 1500 mg in a volume of 60 mL NPO 8 hrs AM bib.
  Interventions: Drug: Nezavist SDD
- Nezavist Cohort 3 (Experimental): Nezavist 4500 mg in a volume of 60 mL NPO 8 hrs AM bib.
  Interventions: Drug: Nezavist SDD
- Nezavist Cohort 4 (Experimental): Nezavist 13500 mg in a volume of 60 mL NPO 8 hrs AM bib.
  Interventions: Drug: Nezavist SDD
- Placebo (Placebo Comparator): Placebo to match 5.4 g of Avicel in a volume of 60 mL NPO 8 hrs AM bib.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nezavist SDD — Formulated as a spray dried dispersion (SDD) suspended in a flavored diluent.
  Other Names: DCUK-OEt
  Arms: Nezavist Cohort 1; Nezavist Cohort 2; Nezavist Cohort 3; Nezavist Cohort 4
Drug: Placebo — Formulated in a diluent that matches the Nezavist SDD suspension in appearance.
  Other Names: Microcrystalline Cellulose
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine the safety, tolerability and effects of Nezavist in healthy adults. The main questions it aims to answer are:

* What is the safety and maximum tolerated dose (MTD) of orally administered Nezavist formulated as a spray dried dispersion (SDD) in healthy volunteers?
* What are the pharmacokinetics (PK) of orally administered Nezavist SDD and its major metabolite (DCUKA) across a range of doses in healthy volunteers?

Researchers will compare the active drug (Nezavist) and a placebo (an inactive substance that looks like the drug) to see if there is any differences between the two groups to make sure Nezavist is safe to use in future studies for reducing alcohol consumption by individuals that have alcohol use disorder (AUD).

DETAILED DESCRIPTION:
Eligible participants will undergo intake procedures and baseline evaluations at the clinic the day before dosing. The next day, participants will be randomized to, and receive, either Nezavist SDD oral suspension or placebo vehicle (4 cohorts of escalating doses of Nezavist with 6 Nezavist subjects and 2 placebo subjects in each cohort). Participants will remain in the clinic for at least an additional 48-hours for safety assessments and blood collections to determine plasma levels of Nezavist, then will be discharged from the clinic and return for follow-up safety tests 72-hours later.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteer, aged 18-to-55 years-of-age, inclusive.
2. BMI must be between 18 and 32 kg/m^2 (inclusive) and weigh a minimum of 50 kg (110 lbs). BMI is calculated as weight in kg divided by the square of height measured in meters.
3. A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG) at the screening visit.
4. If female, be postmenopausal (at least 2 years prior to dosing) or agree to use an acceptable form of birth control from screening until 1 week after dosing. Subjects who claim postmenopausal status will have status confirmed with a follicle stimulating hormone (FSH) test. Acceptable forms of birth control for females include the following:

   * Vasectomized partner (at least 6 months prior to dosing)
   * Surgical sterilization (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) at least 6 months prior to dosing
   * Non-surgical permanent sterilization (eg, Essure procedure) at least 3 months prior to dosing.
   * Double barrier (diaphragm with spermicide; condoms with spermicide)
   * Non-hormonal containing intrauterine device (IUD)
   * Abstinence (must agree to use a double barrier method if they become sexually active during the study)
5. If male, agree to use an acceptable method of birth control during the study and in the 1 week following dosing. Acceptable forms of birth control for males include the following:

   * Vasectomy (at least 6 months before dosing)
   * Partner is surgically sterilized (see methods above for females)
   * Partner uses oral, injectable, or implantable hormonal contraceptives or IUD
   * Double barrier (partner uses diaphragm with spermicide; condoms with spermicide)
   * Abstinence (subject must agree to use a double barrier method if subject becomes sexually active during the study)
6. Be able to verbalize an understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English.
7. Complete all assessments required at screening and baseline and be available to stay in the Phase I unit for a period of approximately 4-days and return for follow-up visits.
8. Be someone who in the opinion of the investigator would be expected to complete the study protocol.

Exclusion Criteria:

1. History of significant sensitivity to any drug.
2. Requirement for any over-the-counter and/or prescription medication, vitamins and/or herbal supplements on a regular basis or use of any of the above within the 2 weeks or 5 half-lives of the respective medication prior to study drug administration.
3. Not have reported taken any medications known to cause significant GI toxicity.
4. More than moderate alcohol consumption in the past 8 weeks. Moderate alcohol consumption is defined as limiting intake to 2 drinks or less in a day for men and 1 drink or less per day for women. Examples of one drink include: Beer: 12 fluid ounces (355 milliliters); Wine: 5 fluid ounces (148 milliliters); Distilled spirits (80 proof): 1.5 fluid ounces (44 milliliters)
5. Have a urine toxicology screen positive during screening or baseline for any of the following substances:

   1. benzodiazepines,
   2. cocaine,
   3. opioids,
   4. amphetamines,
   5. buprenorphine,
   6. methadone,
   7. methamphetamines
   8. oxycodone,
   9. tetrahydrocannabinol (THC)
   10. MDMA
   11. Barbiturates
   12. ethyl glucuronide for recent alcohol use
6. If female, positive pregnancy test or nursing.
7. Positive test result for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab).
8. Positive SARS-CoV-2 antigen test within 72-hours prior to clinic intake.
9. Suspected or known history of Human Immunodeficiency Virus (HIV).
10. History of any clinically significant cardiac, respiratory (except mild asthma), renal, hepatic, GI, hematologic, endocrine, dermatological, metabolic, neurological (nerve injury) or psychiatric disease or disorder, or any uncontrolled medical illness.
11. History of gastric ulcers or known gastric sensitivity to non-steroidal anti-inflammatory drugs.
12. Current symptoms of gastritis or potential GI ulcer complications or screening FOBT positive for blood in the stool.
13. History of head trauma with loss of consciousness, history of epilepsy, seizures or convulsions, including febrile, alcohol or drug withdrawal seizures.
14. Use of any known strong CYP3A4 inhibitors (e.g., ketoconazole) or dual CYP3A4 and 2C9 inhibitor (eg. fluconazole), or dual CYP3A4 and 2C9 inducer (eg. rifampin), or use of any monoamine oxidase inhibitors (MAOIs) within 1 month prior to study drug administration.
15. A clinically notable vital sign abnormality including a history of syncopal or near syncopal events following abrupt change in posture.
16. Have any of the following at screening or baseline:

    * Blood pressure: systolic greater than140 mmHg, diastolic greater than 90 mmHg at Screening or Day -1.
    * Heart rate: greater than 100 beats/minute at screening or Day -1
17. Has a clinically significant laboratory test that is greater than 20% of the upper and lower limit of normal. An out of range normal limit laboratory value is clinically significant if associated with one of the following: a) clinical diagnosis; b) systemic signs and symptoms; or c) physical exam finding.
18. History of cardiac disease, including family history of long-QT syndrome, second degree heart block Type II, third degree heart block or unexplained sudden deaths in their family.
19. Has a clinically significant abnormal ECG or an ECG with a QTc interval corrected for heart rate using the Fridericia formula (QTcF) greater than 430 msec.
20. History of gastric surgery, vagotomy, bowel resection or any surgical procedure that might interfere with GI motility, pH or absorption.
21. Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration.
22. Receipt of any investigational product within 6 weeks prior to study drug administration.
23. Consumption of alcohol within the 1-day period prior to study drug administration
24. Consumption of grapefruit or grapefruit products from 3 days prior to study drug administration to study drug administration.
25. Use of tobacco or nicotine-containing products within the 6-month period preceding study drug administration.
26. Current enrollment in another clinical study.
27. Previous enrollment in this study resulting in administration of nezavist or placebo.
28. Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive nezavist.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety, as measured by the severity, frequency, and relationship of adverse events (AEs) in participants | Serious AEs from the time of informed consent (all other AEs from dosing) through to the follow up visit, up to 7 days, unless serious or if the study physician assesses them to be clinically significant
  Safety is assessed by collecting AEs, including changes from baseline of vital signs, physical examinations, electrocardiograms, fecal occult blood tests, gastrointestinal symptoms and stool consistency, Profile of Moods State (POMS), and clinical laboratory tests (chemistry, hematology, coagulation tests, pregnancy tests, and urinalysis). AEs will be assessed daily after the start of dosing, with closer evaluations in the 12-hour period after the start of dosing
Maximum Tolerated Dose (MTD) of Nezavist in healthy volunteers | From dosing through to the follow up visit, up to 7 days
  The MTD is considered the highest dose where no participants who receive active study drug met the study stopping criteria

SECONDARY OUTCOMES:
Pharmacokinetics AUC-t | From predose through clinic release on Day 3
  Area under the plasma concentration-time curve from time 0 to the time (t) of last quantifiable concentration (Ct) calculated by the log-linear trapezoidal rule
Pharmacokinetics AUC-infinity | From predose through clinic release on Day 3
  Area under the plasma concentration-time curve from time 0 extrapolated to infinity. The terminal area from Ct to infinity is calculated by using the approximation as Ct/λz thus AUC∞ = AUCt + Ct/λz
Pharmacokinetics Cmax | From predose through clinic release on Day 3
  The maximum observed plasma concentration
Pharmacokinetics tmax | From predose through clinic release on Day 3
  The observed time to reach the maximum plasma concentration
Pharmacokinetics λz | From predose through clinic release on Day 3
  The terminal-phase exponential rate constant as calculated from the negative slope of the regression line for the terminal linear portion of the natural log (ln) transformed plasma concentration versus time curve
Pharmacokinetics t1/2 | From predose through clinic release on Day 3
  The apparent terminal exponential half-life, calculated as ln(2)/λz

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wallace, MD, Principal Investigator — University of California, San Diego
Locations (1):
- The Altman Clinical and Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No